CLINICAL TRIAL: NCT05220046
Title: An Exploratory Pilot Study of Palliadelic Treatment to Reduce Psychological Distress in People With Pancreatobiliary and Other Advanced Gastrointestinal Cancers
Brief Title: Palliadelic Treatment to Reduce Psychological Distress in Persons With Advanced Gastrointestinal Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Nebraska University Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0860-21-FB
Record Dates: First submitted 2022-01-15; First posted 2022-02-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pancreas Cancer; Biliary Tract Cancer; Psychological Distress; Gastrointestinal Cancer
Keywords: inoperable; unresectable; stage IV
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Gastrointestinal Neoplasms | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Participants are enrolled as patient/family dyad, with patient in intervention arm and family in observational arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin Treatment Arm (Experimental): Participant with pancreatobilliary cancer will receive 25mg of psilocybin in one 8-hour monitored session with supportive counseling before and after session.
  Interventions: Drug: Psilocybin
- Family Observation Group (No Intervention): The study participant will select a family member who will provide parallel data regarding distress related to pancreatobiliary cancer.

INTERVENTIONS:
Drug: Psilocybin — Psilocybin, 25mg administered orally drug during an 8-hour monitored session with supportive pre- and post- session counseling
  Other Names: mushroom
  Arms: Psilocybin Treatment Arm

SUMMARY:
The primary objective of this study is to evaluate the ability to recruit and retain participants, and to successfully conduct a psilocybin-based protocol, for a study of the treatment of distress related to stage IV or inoperable gastrointestinal cancers. Secondary objectives include pre/post, and longitudinal measurement of distress in intervention participants and a paired family member who is in an observational arm.

DETAILED DESCRIPTION:
Participants with stage IV or inoperable gastrointestinal cancers are eligible for intervention, paired family member recruited for observational arm. Following preparatory sessions in outpatient palliative care clinic or by telehealth (2-4 sessions lasting 60-90 minutes each), psilocybin will be administered as a 25mg capsule during an 8-hour monitored session. Integration sessions (2-3 sessions lasting up to 90 minutes each) will take place in the outpatient palliative care clinic or by phone or tele-heath. Primary and secondary objectives are complete at one-week post treatment, longitudinal exploratory measures collected up to 12 months post baseline.

Parallel assessment of health care utilization, including choices regarding anti-cancer treatment and resource utilization, and family member distress, family communication, well-being and bereavement will be conducted at concurrent time points.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 19 and 85
* Has stage IV or unresectable GI malignancy
* Resides within a 170-mile radius of Omaha, NE
* Speaks English
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Life expectancy ≥ 8 weeks as determined by referring oncologist
* Ability to provide written informed consent and comply with study procedures
* Awareness of the neoplastic and likely incurable nature of his/her disease
* Has one family member willing to participate in measures
* Agreeable to using an adequate method of contraception or birth control from the time of enrollment to 24 hours following the psilocybin session (male and female participant of childbearing potential, defined as age <55 and menses within the prior 2 years with intact ovaries and uterus)
* Negative pregnancy test result (female participants)

Exclusion Criteria:

* Long-term or unstable psychiatric illness that would prevent safe cessation of psychotropic drugs including MAOIs, lithium, or anti-psychotics
* Severe symptoms of depression or anxiety warranting immediate impatient evaluation or treatment
* High-risk of suicide, as measured by Columbia Suicide Severity rating Scale
* Current or prior history of schizophrenia, psychotic disorder (unless substance induced or due to medical condition) or bipolar I or II disorder
* First-degree family member with schizophrenia, psychotic disorder (unless substance induced or due to medical condition) or bipolar I or II disorder
* Conditions known to be incompatible with establishment of rapport or safe exposure to psilocybin including dissociative disorder, borderline personality, traumatic brain injury, obsessive compulsive disorder, anorexia nervosa, or bulimia nervosa
* Alcohol or recreational drug abuse disorder, excluding caffeine and nicotine
* Known CNS metastases or other major CNS disease such as seizure disorder, dementia, Parkinson's disease, multiple sclerosis
* Receive treatment in another clinical trial involving an investigational product for the treatment of cancer during the interventional stage of the protocol
* Advanced hepatic dysfunction as indicated by a Child-Pugh Score of C
* Renal dysfunction as indicated by creatinine clearance <40 ml/min using the Cockroft-Gault equation
* Cardiac or circulatory dysfunction defined as uncontrolled hypertension (systolic blood pressure > 140 or diastolic blood pressure >90 mmHg on three separate readings), angina, stroke or myocardial infarction in the prior 6 months, or claudication
* History of seizures
* Unable to skip a meal (lunch), or have diabetes which requires administration of medication more than twice daily, or with symptomatic hypoglycemia within the prior 30 days
* Pregnant or breastfeeding
* Currently using any of the following potent metabolic inducers or inhibitors

  * Inducers: rifampin, rifabutin, rifapentine, carbamazepine, phenytoin, phenobarbital, nevirapine, efavirenz, St. Johns Wort, or Paclitaxel and dexamethasone (latter two permitted if 5 half-lives have passed between last dose and psilocybin session)
  * Inhibitors: All HIV protease inhibitors, itraconazole, ketoconazole, erythromycin, clarithromycin, troleandomycin
* Metal in body (i.e. hearing aid, cardiac pacemaker, bone plates, braces, non-removeable piercings/implants, etc.) claustrophobia, inability to lay still for one-hour, or any other condition that would preclude MRI scanning

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 18 months
  Number of participants enrolled/ number approached.
Retention Rate | 24 months
  Number of participants who complete the psilocybin session and the assessments at 8-12 days post-psilocybin session/ total enrolled

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) Depression Scale total score from Baseline to 1 week post-dose | Baseline; Day 8-11 post-dose
  Patient Health Questionnaire-9 (PHQ-9) is a nine-item, 32 point scale of frequency of common depressive symptoms. Higher score indicates worse depression.
Change in General Anxiety DIsorder-7 (GAD-7) total score from Baseline to 1 week post-dose | Baseline; Day 8-11 post-dose
  Change in General Anxiety DIsorder-7 (GAD-7) is a 7 item, 21 scale to measure frequency of common symptoms of anxiety with higher score indicating higher severity.
Change in Demoralization Scale (D-II) total score from Baseline to 1 week post-dose | Baseline; Day 8-11 post-dose
  Change in Demoralization Scale (D-II) is a 16 item, 32 point scale with two factors, meaning & purpose and distress & coping, that measures frequency of symptoms of demoralization and existential distress, with higher score indicating higher severity.

CONTACTS AND LOCATIONS:
Overall Officials: Lou Lukas, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No